CLINICAL TRIAL: NCT04686695
Title: Transcutaneous Auricular Vagus Nerve Stimulation for the Treatment of Meniere Disease: a Pilot Study
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation Treatment on Meniere Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: taVNS-MD-2020
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2020-12

CONDITIONS: Meniere Disease
Keywords: Transcutaneous auricular vagus nerve stimulation
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous Auricular Vagus Nerve Stimulation (Experimental)
  Interventions: Device: taVNS

INTERVENTIONS:
Device: taVNS — taVNS was applied using a Huatuo stimulator (SDZ-IIB) developed by Suzhou manufacture of Medical Device and Material. Stimulation parameters was 1 mA of electrical current at a frequency of 20 Hz with pulse duration ≤ 1 ms, for 30min,administered twice daily.

SUMMARY:
Objective: To evaluate the effect of Transcutaneous auricular vagus nerve stimulation for the patients Meniere disease.

Methods: We accrued 25 patients at Beijing TongRen Hospital. All treatments were self-administered by the patients at home after training at the hospital. Patients completed questionnaires at baseline and after 4 weeks, 8 weeks, 12 weeks.

Tinnitus Handicap Inventory (THI), Dizziness Handicap Inventory (DHI), Pure Tone Audiometry, visual scale of ear stuffiness and SF-36 were performed to evaluate the therapeutic effects.

A difference of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 and Age <=70.
2. Clinical diagnosis of meniere disease.

Exclusion Criteria:

1. History of depression, tumors, thyroid disease, diabetes, cardiac diseases.
2. History of Otorhinolaryngology surgery.
3. Pregnant or lactating women.

Ages: 40 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline in the Tinnitus Handicap Inventory (THI) rating scale at 12 Weeks | Day 0 and postintervention at Week 12
  Tinnitus Handicap Inventory (THI) to measure the subjective tinnitus symptoms. Tinnitus Handicap Inventory (THI) to measure the subjective tinnitus symptoms
Mean change from Baseline in the Dizziness Handicap Inventory (DHI) at 12 Weeks | Day 0 and postintervention at Week 12
  DHI to measure the subjective dizziness symptoms.
Mean change from Baseline in the Pure Tone Audiometry at 12 Weeks | Day 0 and postintervention at Week 12
  Pure Tone Audiometry to measure the audition.

SECONDARY OUTCOMES:
Mean change from Baseline in the 36-items Short Form(SF-36) at 12 Weeks | Day 0 and postintervention at Week 12
  SF-36 to measure quality of life
Mean change from Baseline in the visual scale of ear stuffiness at 12 Weeks | Day 0 and postintervention at Week 12
  Visual scale to measure the subjective ear stuffiness symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China